CLINICAL TRIAL: NCT05460663
Title: Improving Resiliency in U.S. Air Force Healthcare Personnel
Brief Title: Improving Resiliency in Air Force Personnel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Stephen H. Hernandez, Associate Professor, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FWR20200166E; N20A19IR (Other Grant/Funding Number: TriService Nursing Research Program); HRRC 20-522 (Other: University of New Mexico Health Science Center HRRC)
Record Dates: First submitted 2022-07-07; First posted 2022-07-15 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Military Personnel; Health Promotion
Keywords: Air Force; Military; Stress; Resilience

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-person SMART training (Experimental): The two-hour VTC or in-person will be provided SMART synchronously to a maximum of 10 individuals. A study team member will contact participants in the VTC group to provide available dates and times of scheduled classes, and these participants will be scheduled for a class they would like to attend. Participants in the VTC group will be provided a web-link prior to the session, and each session will have a unique password to access the training. Participants in the on-line training group will be provided a code to access the training website. If local conditions permit in-person group meetings (i.e. Health Protection Condition [HPCON] Alpha or Bravo), in-person group SMART training in a classroom will be offered as an alternative to VTC sessions. VTC and in-person sessions were provided using the same materials and methods, with the same instructors. Therefore, these are considered to be 'In-Person".
  Interventions: Behavioral: Stress Management and Resilience Training (SMART)
- CBT SMART training (Experimental): SMART will be provided via completion of a self-paced, on-line version completed over a period of four to eight weeks.
  Interventions: Behavioral: Stress Management and Resilience Training (SMART)

INTERVENTIONS:
Behavioral: Stress Management and Resilience Training (SMART) — The Stress Management and Resilience Training (SMART) program was developed by Dr. Amit Sood. SMART focuses on improving the practices of gratitude, mindful presence, kindness, and developing a resilient mindset. The SMART program incorporates practices that focus on six individual factors that have been found to promote individual-level resilience: positive coping, positive affect, positive thinking, realism, behavioral control, and altruism. In this proposed study, SMART will be provided via either a two-hour, video teleconference (VTC) and in-person training or by completion of a self-paced, on-line version completed over a period of four to eight weeks.

SUMMARY:
The study purpose is to examine the effectiveness of the Stress Management and Resilience Training (SMART) in increasing resilience in Air Force (AF) healthcare personnel. SMART includes practices that focus on six factors that promote individual-level resilience. A pretest-posttest, randomized control trial will be used to examine the effectiveness of SMART and is guided by the Defense Centers of Excellence Resilience Continuum. After institutional review board approval, the principal investigator (PI) will recruit a sample of AF healthcare personnel assigned to the 88th Medical Group or USAF School of Aerospace Medicine at Wright Patterson AF Base.

SMART will be provided via either a two-hour, video teleconference (VTC) or in-person training or a self-paced, on-line version completed over four to eight weeks. VTC or on-line versions will be utilized to prevent transmission of COVID-19. If in-person training is feasible and safe at a future point in time, in-person training will replace VTC training.

A baseline survey will include questions regarding age, gender, marital status, race, ethnicity, previous deployment, military rank, and military job duty. The Connor Davidson 10-Item Resilience Scale has demonstrated reliability and validity, and has been used in studies to measure service member resilience. Additional measures include the Perceived Stress Scale, Generalized Anxiety Disorder Scale, and a Quality of Life measure. The CD-10, PSS, GAD-7, and QoL measure will be readministered 12, 18, and 24-weeks after SMART completion.

Initial analysis will include descriptive statistics to characterize demographics, military grade, duty location, and previous deployment status. Cronbach's α will be calculated for each scale. Analyses will be reported as point estimates with 95% confidence intervals and estimates of effect size. Both VTC and on-line groups will be analyzed separately and scores will be pooled to test for overall intervention effects.

Regression models will be conducted on the pre-post intervention difference while controlling for demographic characteristics and previous deployment. The investigators will consider clustering effects among participants from the same organizational unit using random effects. Changes in resilience, stress, anxiety, and QoL over time will be assessed by analyzing changes from baseline to weeks 12, 18, and 24. The investigators will consider a joint analysis of resilience, stress, anxiety, or QOL.

DETAILED DESCRIPTION:
A pre/post-training randomized control trial is proposed to examine the effectiveness of the Stress Management and Resilience Training in increasing the levels of resiliency in healthcare personnel serving in the U.S. Air Force.

Intervention Group Assignment. Simple randomization will be utilized for participant assignment into the intervention delivery type (i.e. VTC/in-person group sessions or on-line SMART program). However, participants will be allowed to switch to their desired delivery type. The investigators will track those individuals who chose to switch their randomized assignment. If in-person training becomes feasible and safe during the planned study period, in-person training will be used to supplement or replace VTC. VTC and in-person sessions are provided using the same materials and methods, with the same instructors. Therefore, these are considered to be 'In-Person". Based on our estimation of the sample size needed and potential attrition, the investigators will seek to enroll at least 60 participants into both the VTC and on-line training groups.

The investigators will assess the participants' level of resilience at baseline (enrollment) and at 12, 18, and 24 weeks post SMART training. A second post-test will be attempted for participants who completed the SMART training no later than the end of February 2021 to test for longer-term changes in resilience.

Sample Size. The investigators have conducted a thorough analysis to determine a sample size for this proposed study using information derived from the available literature. The investigators considered changes in CD-RISC scores, the primary outcome, from baseline to 12 weeks post-intervention after receiving SMART training (efficacy). Assuming a pre-post intervention change in CD-RISC scores of 7.7 (SD = 8.7) to be achievable and meaningful. This corresponds to a standardized mean difference between 0.8 and 0.9 SD. Sample size estimates specified a two-tailed alpha error of .05 for either paired or two-sample t-tests or corresponding nonparametric tests (i.e. Wilcoxon signed ranks or rank sum tests) using a range of effect size and power specifications for mean difference.

Based on this analysis, the investigators propose to recruit 120 active duty service members in total. Assuming up to 25% attrition between enrollment and 12 weeks post-intervention follow-up (i.e. a final sample of 90 or 45 per group), this would be sufficient to achieve 90% power to detect a standardized mean difference of 0.5 SD in either a paired t-test or Wilcoxon signed ranks test.

Intervention. SMART is focused on improving the practices of gratitude, mindful presence, kindness, and developing a resilient mindset. In this study, SMART will be offered via a two-hour VTC training provided by the PI or a qualified AI or via a self-paced on-line course. The two-hour VTC will be provided synchronously to a maximum of 10 individuals. A study team member will contact participants in the VTC group to provide available dates and times of scheduled classes, and these participants will be scheduled for a class participant would like to attend. Participants in the VTC group will be provided a web-link prior to the session, and each session will have a unique password to access the training. Participants in the on-line training group will be provided a code to access the training website. If local conditions permit in-person group meetings (i.e. Health Protection Condition [HPCON] Alpha or Bravo), in-person group SMART training in a classroom will be offered as an alternative to VTC sessions.

In order to provide the in-person or VTC SMART training, instructors must complete the Transform course in Rochester, MN or at another designated location. The Transform course consists of two days of initial classroom training, at least three months of distance-learning with the developer of the SMART training, and a one-day, end-of-course classroom training.

At the end of the course, participants will be offered a copy of SMART with Dr. Sood: The Four-Module Stress Management and Resilience Training Program at no charge to the participants. This book will serve as a review of the practices and course content for improving gratitude, mindful presence, kindness, and developing a resilient mindset. Additionally, in previous studies, individual participants were contacted by phone four weeks after attending the SMART course. These phone calls were offered to provide participants the opportunity to ask questions and to provide reinforcement of the principles presented during the SMART training. Therefore, study participants will be contacted by the PI two weeks after completing the SMART training by e-mail or phone and asked if participants would like to schedule a follow-up phone meeting. If so, the PI will work to schedule a 30-minute follow-up phone call with participants. At the end of this follow-up session, participants will be provided the option to schedule a final 30-minute follow-up phone call. All phone consultations will be completed before the 12-week follow-up survey. These consultations will be a budget item for the proposed study and provided at no cost to participants.

Procedures. Letters of support have been received from the 88th MDG and USAFA Commanders. These letters of support includes permission to recruit potential participants with posted flyers, newspapers, social media, and informational e-mail announcements. Recruitment materials will be distributed in accordance with any limitations set by the governing IRBs and any future Commander instructions. Study information will be distributed as broadly as possible.

Initial recruitment and randomization will be completed during months 3 through 10 of the study. However, if the study team determines the need to recruit additional participants to ensure adequate statistical power, additional participants will be recruited in month 11 and 12. The study team will work with identified local points of contact to develop a schedule to assure the maximum number of participants can receive information about SMART during a variety of times. If approved by the chain of command, SMART could be completed during the participants' scheduled period of work.

After informed consent is obtained and prior to the delivery of the intervention, a survey will be administered to collect demographic information and baseline measurements with the CD-RISC, PSS, GAD-7, and QoL measures. Participant demographic data, e-mail and phone contact information, and responses to survey items will be initially completed using a paper survey prior to the delivery of SMART and manually entered into the Research Electronic Data Capture System (REDCap; DHHS/NIH/NCRR #8UL1TR000041) by a study team member. If a participant prefers, participants will be provided a web-link to enter the initial information directly into REDCap. REDCap is a secure and encrypted, web-based platform licensed to and managed by the University of New Mexico Health Sciences Center Clinical and Translational Science Center (UNM HSC CTSC). REDCap includes a suite of research tools for project management, survey administration, encrypted database storage and retrieval, and reporting. REDCap will be utilized to administer follow-up surveys at week 12, 18 and 24 (if applicable) after participants complete SMART. The investigators propose to collect the 24-week follow-up survey responses in order to conduct an exploratory analysis to assess the longevity of the effect of SMART on resilience and stress.

Study team members will verify participant data has been entered correctly. Participant e-mail and phone contact information will be used to schedule a follow-up phone call two weeks after completing the SMART training (see intervention). Participants' e-mail contact information will be used be utilized to send follow-up surveys through REDCap. Each survey will take approximately 10 to 15 minutes for participants to complete. If the participant does not respond to the initial REDCap invitation, a maximum of three e-mail reminders (one reminder per week after the initial e-mail is sent) will be sent to complete the survey. If a participant does not complete the survey after all e-mail requests have been sent, a study team member may call the participant to verify their e-mail information and offer to assist the participant with accessing the survey. Because participants' demographic information will be associated with an individual's contact information in REDCap, demographic information will not be requested as part of the surveys at weeks 12, 18 or 24. All data will be de-identified prior to exporting the data for analysis.

Data Analysis. IBM® SPSS® Statistics and R will be used for the statistical analysis. Initial analysis will include descriptive statistics, including means or medians, frequencies and percentages, as appropriate, to characterize demographic status, military grade, duty location, military occupation, and previous deployment status. Cronbach's α will be calculated for each multi-item scale.

The objectives of our analysis include testing and estimating the efficacy of the intervention by comparing pre-post intervention changes (improvements) in the outcome measurements of interest. Analyses will be reported as point estimates with 95% confidence intervals and appropriate estimates of effect size. In this analysis, both the VTC and on-line groups will be analyzed separately and scores will also be pooled together to test for overall intervention effects.

To better understand factors that can impact the intervention effects, the investigators will conduct regression models on the pre-post intervention difference while controlling for demographic characteristics, AFSC, and previous deployment. The investigators will also take into consideration potential clustering effects among the participants from the same organizational unit using random effects (e.g. in regression models).

Changes in resilience, stress, anxiety, and QoL over time will be assessed by separately analyzing changes from baseline to week 12 and to week 24. A joint analysis of the longitudinal trend over the three time points at baseline, 12-week, and 24-week will be completed. The investigators will also consider a joint analysis of resilience, stress, anxiety, or QOL, as well as, analysis for subscales of any specific domain of interest.

Recruitment Plan. Study team members will work to recruit a sample of active component Air Force healthcare personnel. For in-person recruitment sessions, all infection control practices and guidelines required by the installation will be enforced. Informational sessions will be coordinated at the 88th MDG and USAFA to occur at unit or staff meetings and open sessions in prearranged locations. The location, number, and timing of these sessions will be designed to make information about the study accessible to service members on all shifts. Team members will be attired in civilian clothing during these meetings. Informed consent will be completed by a study team member after the completion of the described information sessions with individuals or groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be active component healthcare personnel (any 4XXX Officer or Enlisted AFSC) serving in the U.S. Air Force, assigned to 88th MDG and USAFA at WPAFB, OH.
* Participants must be ≥ 18 years of age to participate.

Exclusion Criteria:

* Adults unable or unwilling to provide consent and individuals who are not yet adults will be excluded from this study.
* Active component Air Force service members without a healthcare AFSC will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Hernandez, PhD, RN, Principal Investigator — University of New Mexico College of Nursing
Locations (1):
- Wright-Patterson Air Force Base, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Meredith LS, Sherbourne CD, Gaillot SJ, Hansell L, Ritschard HV, Parker AM, Wrenn G. Promoting Psychological Resilience in the U.S. Military. Rand Health Q. 2011 Jun 1;1(2):2. eCollection 2011 Summer. PMID 28083176
- [Background] Thompson SR, Dobbins S. The Applicability of Resilience Training to the Mitigation of Trauma-Related Mental Illness in Military Personnel [Formula: see text]. J Am Psychiatr Nurses Assoc. 2018 Jan/Feb;24(1):23-34. doi: 10.1177/1078390317739957. Epub 2017 Nov 15. PMID 29139325
- [Background] Rocklein Kemplin K, Paun O, Godbee DC, Brandon JW. Resilience and Suicide in Special Operations Forces: State of the Science via Integrative Review. J Spec Oper Med. 2019 Summer;19(2):57-66. doi: 10.55460/BQES-AM8H. PMID 31201752
- [Background] Committee on the Assessment of Resiliency and Prevention Programs for Mental and Behavioral Health in Service Members and Their Families; Board on the Health of Select Populations; Institute of Medicine; Denning LA, Meisnere M, Warner KE, editors. Preventing Psychological Disorders in Service Members and Their Families: An Assessment of Programs. Washington (DC): National Academies Press (US); 2014 Feb 11. Available from http://www.ncbi.nlm.nih.gov/books/NBK222170/ PMID 25057692
- [Background] 5 Department of Defense. (2015, July). Report to Congressional Armed Services Committees: Implementation of recommendations of Institute of Medicine on improvements on certain resilience and prevention programs of the Department of Defense. Retrieved from https://www.pdhealth.mil/report-implementation-recommendations-institute-medicine-improvements-certain-resilience-and
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Background] Windle G. The contribution of resilience to healthy ageing. Perspect Public Health. 2012 Jul;132(4):159-60. doi: 10.1177/1757913912449572. No abstract available. PMID 22729003
- [Background] Resilient Option. (n.d.). Resilient option on-line program. Retrieved June 30, 2020 from https://www.resilientoption.com/online-program
- [Background] Loprinzi CE, Prasad K, Schroeder DR, Sood A. Stress Management and Resilience Training (SMART) program to decrease stress and enhance resilience among breast cancer survivors: a pilot randomized clinical trial. Clin Breast Cancer. 2011 Dec;11(6):364-8. doi: 10.1016/j.clbc.2011.06.008. Epub 2011 Aug 10. PMID 21831722
- [Background] Sood A, Prasad K, Schroeder D, Varkey P. Stress management and resilience training among Department of Medicine faculty: a pilot randomized clinical trial. J Gen Intern Med. 2011 Aug;26(8):858-61. doi: 10.1007/s11606-011-1640-x. Epub 2011 Jan 29. PMID 21279454
- [Background] Sood A, Sharma V, Schroeder DR, Gorman B. Stress Management and Resiliency Training (SMART) program among Department of Radiology faculty: a pilot randomized clinical trial. Explore (NY). 2014 Nov-Dec;10(6):358-63. doi: 10.1016/j.explore.2014.08.002. Epub 2014 Aug 21. PMID 25443423
- [Background] Chesak SS, Bhagra A, Schroeder DR, Foy DA, Cutshall SM, Sood A. Enhancing resilience among new nurses: feasibility and efficacy of a pilot intervention. Ochsner J. 2015 Spring;15(1):38-44. PMID 25829879
- [Background] Magtibay DL, Chesak SS, Coughlin K, Sood A. Decreasing Stress and Burnout in Nurses: Efficacy of Blended Learning With Stress Management and Resilience Training Program. J Nurs Adm. 2017 Jul/Aug;47(7-8):391-395. doi: 10.1097/NNA.0000000000000501. PMID 28727625
- [Background] Kashani K, Carrera P, De Moraes AG, Sood A, Onigkeit JA, Ramar K. Stress and burnout among critical care fellows: preliminary evaluation of an educational intervention. Med Educ Online. 2015 Jul 23;20:27840. doi: 10.3402/meo.v20.27840. eCollection 2015. PMID 26208706
- [Background] Stonnington CM, Darby B, Santucci A, Mulligan P, Pathuis P, Cuc A, Hentz JG, Zhang N, Mulligan D, Sood A. A resilience intervention involving mindfulness training for transplant patients and their caregivers. Clin Transplant. 2016 Nov;30(11):1466-1472. doi: 10.1111/ctr.12841. Epub 2016 Oct 14. PMID 27618687
- [Background] Werneburg BL, Jenkins SM, Friend JL, Berkland BE, Clark MM, Rosedahl JK, Preston HR, Daniels DC, Riley BA, Olsen KD, Sood A. Improving Resiliency in Healthcare Employees. Am J Health Behav. 2018 Jan 1;42(1):39-50. doi: 10.5993/AJHB.42.1.4. PMID 29320337
- [Background] Dyrbye LN, Shanafelt TD, Werner L, Sood A, Satele D, Wolanskyj AP. The Impact of a Required Longitudinal Stress Management and Resilience Training Course for First-Year Medical Students. J Gen Intern Med. 2017 Dec;32(12):1309-1314. doi: 10.1007/s11606-017-4171-2. Epub 2017 Aug 31. PMID 28861707
- [Background] Sharma V, Sood A, Prasad K, Loehrer L, Schroeder D, Brent B. Bibliotherapy to decrease stress and anxiety and increase resilience and mindfulness: a pilot trial. Explore (NY). 2014 Jul-Aug;10(4):248-52. doi: 10.1016/j.explore.2014.04.002. Epub 2014 Apr 19. PMID 25037668
- [Background] Bezdjian S, Schneider KG, Burchett D, Baker MT, Garb HN. Resilience in the United States Air Force: Psychometric properties of the Connor-Davidson Resilience Scale (CD-RISC). Psychol Assess. 2017 May;29(5):479-485. doi: 10.1037/pas0000370. Epub 2016 Aug 8. PMID 27504904
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Cohen, S., & Williamson, G. (1988). Perecived stress in a probablility sample of the United States. In S. Spacapan & S. Oskamp (Eds.), The social psychology of health (pp. 31-67). Newbury Park, CA: Sage.
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Locke DE, Decker PA, Sloan JA, Brown PD, Malec JF, Clark MM, Rummans TA, Ballman KV, Schaefer PL, Buckner JC. Validation of single-item linear analog scale assessment of quality of life in neuro-oncology patients. J Pain Symptom Manage. 2007 Dec;34(6):628-38. doi: 10.1016/j.jpainsymman.2007.01.016. Epub 2007 Aug 20. PMID 17703910
- [Background] Hernandez SHA, Morgan BJ, Parshall MB. Treatment-Seeking Beliefs and Behaviors in Air Force Nursing Personnel. Mil Med. 2017 Jul;182(7):e1687-e1692. doi: 10.7205/MILMED-D-16-00397. PMID 28810957
- [Background] Pietrzak RH, Goldstein MB, Malley JC, Rivers AJ, Johnson DC, Southwick SM. Risk and protective factors associated with suicidal ideation in veterans of Operations Enduring Freedom and Iraqi Freedom. J Affect Disord. 2010 Jun;123(1-3):102-7. doi: 10.1016/j.jad.2009.08.001. Epub 2009 Oct 12. PMID 19819559
- [Background] Hernandez SH, Morgan BJ, Parshall MB. Resilience, Stress, Stigma, and Barriers to Mental Healthcare in U.S. Air Force Nursing Personnel. Nurs Res. 2016 Nov/Dec;65(6):481-486. doi: 10.1097/NNR.0000000000000182. PMID 27529539
- [Background] Maguen S, Turcotte DM, Peterson AL, Dremsa TL, Garb HN, McNally RJ, Litz BT. Description of risk and resilience factors among military medical personnel before deployment to Iraq. Mil Med. 2008 Jan;173(1):1-9. doi: 10.7205/milmed.173.1.1. PMID 18251325
- [Background] Sood, A. (n.d.). Transform course. Retrieved June 30, 2020 from https://www.resiliencetrainer.com/transform-course
- [Background] Pietrzak RH, Southwick SM. Psychological resilience in OEF-OIF Veterans: application of a novel classification approach and examination of demographic and psychosocial correlates. J Affect Disord. 2011 Oct;133(3):560-8. doi: 10.1016/j.jad.2011.04.028. Epub 2011 May 31. PMID 21624683
- [Background] Singh JA, Satele D, Pattabasavaiah S, Buckner JC, Sloan JA. Normative data and clinically significant effect sizes for single-item numerical linear analogue self-assessment (LASA) scales. Health Qual Life Outcomes. 2014 Dec 18;12:187. doi: 10.1186/s12955-014-0187-z. PMID 25519478
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Campbell-Sills L, Stein MB. Psychometric analysis and refinement of the Connor-davidson Resilience Scale (CD-RISC): Validation of a 10-item measure of resilience. J Trauma Stress. 2007 Dec;20(6):1019-28. doi: 10.1002/jts.20271. PMID 18157881

RESULTS

PARTICIPANT FLOW:
Groups:
- VTC/In-person SMART Training: The two-hour VTC or in-person will be provided SMART synchronously to a maximum of 10 individuals. A study team member will contact participants in the VTC group to provide available dates and times of scheduled classes, and these participants will be scheduled for a class they would like to attend. Participants in the VTC group will be provided a web-link prior to the session, and each session will have a unique password to access the training. Participants in the on-line training group will be provided a code to access the training website. If local conditions permit in-person group meetings (i.e. Health Protection Condition [HPCON] Alpha or Bravo), in-person group SMART training in a classroom will be offered as an alternative to VTC sessions.
  Stress Management and Resilience Training (SMART): The Stress Management and Resilience Training (SMART) program was developed by Dr. Amit Sood. SMART focuses on improving the practices of gratitude, mindful presence, kindness, and developing a resilient mindset. The SMART program incorporates practices that focus on six individual factors that have been found to promote individual-level resilience: positive coping, positive affect, positive thinking, realism, behavioral control, and altruism. In this proposed study, SMART will be provided via either a two-hour, video teleconference (VTC) or in-person training or by completion of a self-paced, on-line version completed over a period of four to eight weeks.
- CBT SMART Training: SMART will be provided via completion of a self-paced, on-line version completed over a period of four to eight weeks.
  Stress Management and Resilience Training (SMART): The Stress Management and Resilience Training (SMART) program was developed by Dr. Amit Sood. SMART focuses on improving the practices of gratitude, mindful presence, kindness, and developing a resilient mindset. The SMART program incorporates practices that focus on six individual factors that have been found to promote individual-level resilience: positive coping, positive affect, positive thinking, realism, behavioral control, and altruism. In this proposed study, SMART will be provided via either a two-hour, video teleconference (VTC) or in-person training or by completion of a self-paced, on-line version completed over a period of four to eight weeks.
Period: Overall Study
Arm/Group | VTC/In-person SMART Training | CBT SMART Training
Started | 32 | 24
Completed | 30 | 19
Not Completed | 2 | 5
Not completed — Withdrawal by Subject | 2 | 5

BASELINE CHARACTERISTICS:
Population: 56 Completed Baseline Assessment, 49 Completed either in-person/video-teleconference or CBT training. VTC was initially provided due to COVID-19 restrictions. Once these restrictions were reduced, in-person training became feasible. VTC and in-person training was accomplished with the same instructors and materials. Therefore, VTC and in-person training were considered to be equivalent in content and delivery and participants were categorized into one in-person/VTC arm for analysis.
Groups:
- In Person: VTC was initially provided due to COVID-19 isolation and travel restrictions. Once these restrictions were reduced, in-person training became feasible. The VTC and in-person training was accomplished with the same instructors and materials. Therefore, the VTC and in-person training were considered to be indistinguishable and equivalent in content and delivery and participants were categorized into one in-person/VTC arm for analysis.
- Computer Based Training: SMART CBT was provided via completion of a self-paced, on-line version completed over a period of four to eight weeks.
- Total: Total of all reporting groups
Arm/Group | In Person | Computer Based Training | Total
Number analyzed (Participants) | 32 | 24 | 56
Age, Customized [Count of Participants; unit: Participants] — Categorical
  Participants
    <30 years | 7 | 6 | 13
    30+ years | 25 | 18 | 43
Sex: Female, Male [Count of Participants; unit: Participants] — Categorical
  Participants
    Female | 11 | 8 | 19
    Male | 21 | 16 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Categorical
  Participants
    Hispanic or Latino | 3 | 2 | 5
    Not Hispanic or Latino | 28 | 22 | 50
    Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 17 | 15 | 32
  More than one race | 10 | 5 | 15
  Unknown or Not Reported | 0 | 0 | 0
Military Grade [Number; unit: participants]
  Officer | 17 | 11 | 28
  Enlisted | 15 | 13 | 28

OUTCOME MEASURES:

1. Primary Outcome: Changes in Connor-Davidson 10-Item Scale (CD-10)
Description: Resilience was measured using the CD-10, a 10-item scale derived from the original, 25-item Connor Davidson Resilience Scale. Respondents can answer each item using a five-point rating ranging from not true at all (0) to true nearly all the time (4). A total CD-RISC score is calculated by summing the score of all 10 items for a total possible score of 40, with a higher score reflecting a greater level of resilience. The CD-10 has a reported Cronbach's alpha of .85 and has demonstrated construct validity. The scale was administered to each participants at 4 times: baseline, and 12/18/24 weeks after SMART completion.
Time Frame: Changes in self-reported CD-10 from Baseline at 12, 18, and 24 weeks post-SMART completion
Population: Follow-up surveys were voluntary. Up to three reminder surveys were sent at each time point.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- CD-10 (In-Person/VTC): Resilience was measured using the CD-10, a 10-item scale derived from the original, 25-item Connor Davidson Resilience Scale. Respondents answer each item using a five-point rating ranging from not true at all (0) to true nearly all the time (4). A total CD-10 score is calculated by summing the score of all 10 items for a total possible score of 40, with a higher score reflecting a greater level of resilience.
- CD-10 (CBT): CBT
Arm/Group | CD-10 (In-Person/VTC) | CD-10 (CBT)
Number analyzed (Participants) | 32 | 24
score on a scale
  CD-10: Baseline | 28 [25.8 to 32.8] | 28.5 [25.0 to 32.3]
  CD-10: 12 Weeks: number analyzed (Participants) | 18 | 13
  CD-10: 12 Weeks | 33.5 [29.5 to 35.8] | 32 [30 to 33.3]
  CD-10: 18 Weeks: number analyzed (Participants) | 17 | 14
  CD-10: 18 Weeks | 36 [31.1 to 37] | 34 [28.5 to 38]
  CD-10: 24 Weeks: number analyzed (Participants) | 14 | 13
  CD-10: 24 Weeks | 36.5 [30 to 37] | 32.2 [29 to 37]
Statistical Analysis 1: Comparison: CD-10 (In-Person/VTC); Test type: Equivalence — Paired Wilcoxon signed ranks tests were used to compare changes at 12-week, 18-week, or 24-week follow-ups from the baseline scores for all measurements in each training modality separately and combined. Comparisons were made with participants who had data at both baseline and the follow-up. Difference-in-difference comparison of changes between two training modalities at each follow-up from the baseline were made to assess differences between CBT and in-person training; p = .083, Wilcoxon (Mann-Whitney) — The reported P-value is for differences between groups at 24-weeks post-intervention.The Benjamini & Hochberg adjustment was applied to control for the false-discovery rate among all pairwise pre-post comparisons

2. Secondary Outcome: Changes in Perceived Stress Scale (PSS)
Description: The PSS was developed to provide both a global measure and a measure for current levels of perceived stress. The PSS is a 14-item instrument, and respondents answer each item on a four-point scale ranging from never (0) to very often (4). An individual's total score is calculated by reverse scoring seven items and then summing all item scores, resulting in a score range of 0-56, with a higher score reflecting a greater level of stress. The scale was administered to each participants at 4 times: baseline, and 12/18/24 weeks after SMART completion.
Time Frame: Changes in self-reported PSS from Baseline at 12, 18, and 24 weeks post-SMART completion
Population: Follow-up surveys were voluntary. Up to three reminder surveys were sent at each time point.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- PSS Scores (VTC/In-Person): PSS Scores (VTC/In-Person)
- PSS (CBT): CBT
Arm/Group | PSS Scores (VTC/In-Person) | PSS (CBT)
Number analyzed (Participants) | 32 | 24
score on a scale
  Baseline | 24.5 [18.5 to 29] | 24.5 [18.8 to 29.3]
  PSS: 12 Weeks: number analyzed (Participants) | 18 | 13
  PSS: 12 Weeks | 20 [12.5 to 24] | 16 [14 to 21]
  PSS: 18 Weeks: number analyzed (Participants) | 16 | 14
  PSS: 18 Weeks | 16.7 [10.8 to 22.4] | 16.5 [12 to 22.8]
  PSS: 24 Weeks: number analyzed (Participants) | 14 | 24
  PSS: 24 Weeks | 16.5 [12 to 24.8] | 13 [11 to 21]

3. Secondary Outcome: Changes in Generalized Anxiety Disorder Scale (GAD-7)
Description: Anxiety was measured with the GAD-7. Respondents can answer each item using a four-point scale ranging from not at all (0) nearly every day (3). A total score is calculated by summing the scores of the seven items with possible scores ranging from 0-21, with a higher score reflecting a greater level of anxiety. Scores between 5-9 are indicative of mild anxiety, and score between 15-21 are indicative of severe anxiety. The scale was administered to each participants at 4 times: baseline, and 12/18/24 weeks after SMART completion.
Time Frame: Changes in self-reported GAD-7 scores from Baseline at 12, 18, and 24 weeks post-SMART completion
Population: Follow-up surveys were voluntary. Up to three reminder surveys were sent at each time point.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- GAD-7 Scores (In-person/VTC): GAD-7 Scores (In-person/VTC)
- GAD-7 (CBT): GAD-7 CBT
Arm/Group | GAD-7 Scores (In-person/VTC) | GAD-7 (CBT)
Number analyzed (Participants) | 32 | 24
score on a scale
  Baseline | 5.5 [1.8 to 10.3] | 4 [2 to 8.3]
  GAD-7: 12 Weeks: number analyzed (Participants) | 18 | 13
  GAD-7: 12 Weeks | 3 [0.25 to 7.8] | 2 [2 to 6]
  GAD-7: 18 Weeks: number analyzed (Participants) | 16 | 14
  GAD-7: 18 Weeks | 2 [0 to 3.5] | 3 [0 to 5.8]
  GAD-7: 24 Weeks: number analyzed (Participants) | 14 | 13
  GAD-7: 24 Weeks | 2.7 [1.3 to 5.8] | 2 [1 to 7]

4. Secondary Outcome: Changes in Quality of Life (QOL)
Description: A single-item Linear Analogue Self-Assessment (LASA) QoL measure was used to measure overall quality of life for this study. Participants responded to each item using an 11-point Likert scale ranging from as bad as it can be (0) to as good as it can be (10), with a higher score reflecting a greater level of quality of life. The scale was administered to each participants at 4 times: baseline, and 12/18/24 weeks after SMART completion.
Time Frame: Changes in self-reported QOL scores from Baseline at 12, 18, and 24 weeks post-SMART completion
Population: Follow-up surveys were voluntary. Up to three reminder surveys were sent at each time point.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- QoL Scores (In-Person/VTC): QoL Scores (In-Person/VTC)
- QoL Scores (CBT): QoL Scores (CBT)
Arm/Group | QoL Scores (In-Person/VTC) | QoL Scores (CBT)
Number analyzed (Participants) | 32 | 24
score on a scale
  Baseline | 7 [6 to 8] | 8 [7 to 8]
  QoL: 12 Weeks: number analyzed (Participants) | 18 | 13
  QoL: 12 Weeks | 7 [6 to 8.8] | 8 [7 to 8]
  QoL: 18 Weeks: number analyzed (Participants) | 16 | 14
  QoL: 18 Weeks | 8 [6.8 to 8.3] | 7 [7 to 8.8]
  QoL: 24 Weeks: number analyzed (Participants) | 14 | 13
  QoL: 24 Weeks | 8 [7.3 to 8.8] | 7 [7 to 8]

ADVERSE EVENTS:
Time Frame: Participants were recruited over a 9 month period.
Description: 56 participants were monitored for potential risks.
Arm/Group | VTC/In-person SMART Training | CBT SMART Training
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/24
Other Adverse Events (participants affected / at risk) | 0/32 | 0/24

LIMITATIONS AND CAVEATS:
We cannot preclude self-selection bias. Although invitations to participate and reminder e-mails were sent to participants, there was variable completion rates of follow-up surveys. In-person SMART was conducted via VTC and small face-to-face classes. Although the content of face-to-face delivery of SMART was identical to VTC, we do not know if a difference in teaching effectiveness due to the difference in delivery method was present. We were unable to recruit 90 participants, as planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT05460663/Prot_SAP_ICF_000.pdf